CLINICAL TRIAL: NCT07225946
Title: A Phase 3 Randomized, Open-label Study of Pasritamig (JNJ-78278343), a T-cell-redirecting Agent Targeting Human Kallikrein 2, With Docetaxel Versus Docetaxel for Metastatic Castration-resistant Prostate Cancer
Brief Title: A Study of Pasritamig With Docetaxel Versus Docetaxel in Participants With Metastatic Castration-Resistant Prostate Cancer
Acronym: KLK2-PASenger
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78278343PCR3003; 78278343PCR3003 (Other: Janssen Research & Development, LLC); 2025-522713-29-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-11-06; First posted 2025-11-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pasritamig+Docetaxel (Experimental): Participants will receive pasritamig along with docetaxel until the end of trial (EOT) visit or until confirmed radiographic progression by blinded independent central review (BICR), or any other protocol defined criteria are met.
  Interventions: Drug: Pasritamig; Drug: Docetaxel
- Docetaxel (Active Comparator): Participants will receive docetaxel along with prednisone as background medication.
  Interventions: Drug: Docetaxel; Drug: Prednisone

INTERVENTIONS:
Drug: Pasritamig — Pasritamig will be administered.
  Other Names: JNJ-78278343
  Arms: Pasritamig+Docetaxel
Drug: Docetaxel — Docetaxel will be administered.
Drug: Prednisone — Prednisone will be administered.
  Arms: Docetaxel

SUMMARY:
The purpose of this study is to find out whether treatment with pasritamig and docetaxel prolongs radiographic progression free survival (rPFS) (the length of time from start of treatment until disease worsens as determined by scans) when compared to treatment with docetaxel in participants with metastatic castrate-resistant prostate cancer (mCRPC; a cancer of prostate, a male reproductive gland found below the bladder, that grows despite low levels of male hormones).

ELIGIBILITY:
Inclusion criteria:

* Have histologically confirmed adenocarcinoma of the prostate
* Have disease that is metastatic at the time of the screening as determined by the investigator
* Participants must receive ongoing androgen deprivation therapy (ADT) with a gonadotropin releasing hormone (GnRH) analog throughout the treatment or have had prior bilateral orchiectomy, and have serum testosterone less than or equal to (<=) 50 nanogram per milliliter (ng/dL) (<= 1.73 nanomoles per Liter [nmol/L]) at screening
* Have progressed on at least 1 novel androgen receptor pathway inhibition (ARPI) but received no more than 2 different ARPI for any stage of disease. Must have discontinued ARPI before randomization into the study
* Have an eastern cooperative oncology group (ECOG) performance status of 0 to 1

Exclusion criteria:

* Known history of either brain or leptomeningeal prostate cancer metastases
* Participants with known breast cancer gene 1/2 (BRCA 1/2) mutations (germline or somatic) who have not received treatment with a poly (ADP-ribose) polymerase (PARP) inhibitor, unless not available or contraindicated
* Prior or concurrent second malignancy (other than the disease under study) because the natural history or treatment could interfere with study endpoints
* Received cytotoxic chemotherapy for prostate cancer in any setting
* Received prior treatment with human kallikrein 2 (KLK-2) directed therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-11-19 (Estimated); Study Completion 2029-06-20 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS) Assessed by BICR | Up to approximately 1 years 10 months
  rPFS is assessed by BICR and is defined as the time from the date of randomization to the first date of radiographic disease progression, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 4 years 5 months
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Time to Symptomatic Progression (TSP) | Up to approximately 4 years 5 months
  TSP is defined as the time from the date of randomization to the date of the first occurrence of any of the following: the use of external beam radiation for skeletal or pelvic symptoms, the need for tumor-related orthopedic surgical intervention, other cancer-related procedures, cancer-related morbid events, and initiation of a new systemic anticancer therapy because of cancer symptoms.
Time to Subsequent Therapy (TST) | Up to approximately 4 years 5 months
  TST is defined as time from randomization to the initiation of any subsequent systemic anticancer therapy.
Time to Skeletal-Related Event (TSRE) | Up to approximately 4 years 5 months
  TSRE is defined as the time from the date of randomization to the date of first occurrence of any of the following: the use of external beam radiation therapy to relieve skeletal symptoms, the need for tumor-related orthopedic surgical intervention, the occurrence of new bone fractures (cancer-related; vertebral or non-vertebral) or the occurrence of tumor-related spinal cord compression.
Objective Response Rate (ORR) | Up to approximately 4 years 5 months
  ORR is defined as the proportion of participants who have measurable disease at baseline and have complete response (CR) or partial response (PR) or better by objective radiographic disease evaluation per response evaluation criteria in solid tumors (RECIST) version.1.1 response criteria and no bone progression as per prostate cancer working group 3 (PCWG3) as determined by the BICR.
Duration of Response (DOR) | Up to approximately 4 years 5 months
  DOR will be calculated among responders (PR or better) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the PCWG3 or RECIST version 1.1 response criteria, or death due to any cause, whichever occurs first.
Time to Prostate-Specific Antigen (PSA) Progression | Up to approximately 4 years 5 months
  Time to PSA progression will be calculated from date of enrollment to the date of first documentation of PSA progression. As per Prostate Cancer Clinical Trials Working Group (PCWG2) criteria, PSA progression is defined as greater than or equal to (>=) 25 percent (%) and >=2 nanogram/milliliter (ng/mL) after 12 weeks (in case of no decline in PSA from Baseline), or first PSA increase that is >=25% and >=2 ng/mL above the nadir, and which is confirmed by a second value 3 or more weeks later (in case of decline of PSA from baseline).
Proportion of Participants Who Achieved Prostate-Specific Antigen (PSA) 50 Response | Up to approximately 4 years 5 months
  PSA-50 response is defined as the proportion of participants with a reduction in blood concentration of PSA (ng/mL) to 50% from baseline, confirmed by a second value.
Proportion of Participants Who Achieved Prostate-Specific Antigen (PSA) 90 Response | Up to approximately 4 years 5 months
  PSA-90 response is defined as the proportion of participants with a reduction in blood concentration of PSA (ng/mL) to 90% from baseline, confirmed by a second value.
Duration of PSA Response | Baseline and up to approximately 4 years 5 months
  Duration of a PSA response is the time taken to achieve a PSA response that is decrease in PSA from baseline by >= 50%.
Progression Free Survival After Subsequent Therapy (PFS2) | Up to approximately 4 years 5 months
  PFS2 is defined as the time from randomization to the date of progression (radiographic, clinical, or PSA progression) on the first subsequent anti-cancer (second progression), or death from any cause, whichever comes first.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) by Severity | Up to approximately 4 years 5 months
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. An SAE: results in death, is life-threatening, requires inpatient hospitalization or prolonging hospitalization, results in disability, is a congenital birth defect, is a suspected transmission of any infectious agent via a medicinal product, is indicating suicidal ideation, is medically important. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. by using standard grades as follows: Grade 1: Mild; asymptomatic or mild symptoms; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; Grade 3: Severe but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening consequences; and Grade 5: Death related to AE.
Number of Participants With Clinical Laboratory Abnormalities | Up to approximately 4 years 5 months
  Participants with laboratory abnormalities (hematology, serum chemistry, coagulation, and tumor markers) will be reported.
Change from Baseline in Health Related Quality of Life (HRQoL) as Assessed by Brief Pain Inventory-Short Form (BPI-SF) | Baseline up to approximately 4 years 5 months
  The BPI-SF was developed to measure both intensity or severity of pain and pain interference with daily life dimensions. It measures pain intensity via 4 questions, that is, "pain at its worst in the last 24 hours", "pain at its least in the last 24 hours", "
Change from Baseline in HRQoL as Assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Cancer Module (EORTC QLQ-C30) Scale Score | Baseline up to approximately 4 years 5 months
  The EORTC QLQ-C30 - Version 3 is a self-administered, 30-item questionnaire measuring the health-related quality of life of participants with cancer. EORTC QLQ-C30 includes 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), a global health status / quality of life scale, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much". Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent". A high score for a functional scale represents a high level of functioning, whereas a high score for a symptom scale/single item represents a high level of symptom.
Change from Baseline in HRQoL as Assessed by EORTC Quality of Life Questionnaire-Prostate (EORTC QLQ-PR25) Scale Score | Baseline up to approximately 4 years 5 months
  The EORTC QLQ-PR25 is a self-completed instrument was specifically designed for prostate cancer patients and includes 25 items that cover 6 dimensions: (1) PR URI (urinary symptoms, 8 items), (2) PR BOW (bowel symptoms, 4 items), (3) PR HTR (hormonal treatment-related symptoms, 6 items), (4) PR AID (incontinence aid, 1 item), (5) PR SAC (sexually active, 2 items); and (6) PR SFU (sexual function, 4 items). Higher scores on symptom domains (for example., urinary, bowel, etc.) indicate greater symptom burden and higher scores on function domains (for example, Sexual Function) indicate better functioning.
Change from Baseline in HRQoL as Assessed by European Quality of Life Visual Analog Scale (EQ-5D VAS) Score | Baseline up to approximately 4 years 5 months
  The EQ-5D descriptive system comprises 5 items across the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D includes a visual analog scale (EQ-VAS) that has endpoints labeled "best imaginable health state" and "worst imaginable health state" anchored at 100 and 0, respectively. Here, higher score indicates better quality of life.
Time to Sustained Worsening of Pain as Assessed by BPI-SF | Up to approximately 4 years 5 months
  Time to sustained worsening of pain will be reported using BPI-SF. The BPI-SF was developed to measure both intensity or severity of pain and pain interference with daily life dimensions. It measures pain intensity via 4 questions, that is, "pain at its worst in the last 24 hours", "pain at its least in the last 24 hours", "pain on the average", and "pain you have right now". The BPI-SF assesses how much pain has interfered with the following 7 activities: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Higher score indicates more pain.
Treatment Side Effect as Assessed by EORTC IL-6 Score | Up to approximately 4 years 5 months
  The EORTC IL46 is a single question that assesses bother (burden) of treatment. It is rated on a scale from 1 to 4, ranging from "not at all" to "very much"
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) Scale Score | Up to approximately 4 years 5 months
  The EQ-5D descriptive system comprises 5 items across the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L uses a 5-point Likert response scale ranging from "No problems" to "Extreme problems". Here, higher score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- United States (6):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Profound Research LLC at Cancer and Leukemia Center, Sterling Heights, Michigan
  - HealthPartners Frauenshuh Cancer Center CRC West, Saint Louis Park, Minnesota
  - HealthPartners Cancer Center at Regions Hospital CRC East, Saint Paul, Minnesota
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Houston Metro Urology, Houston, Texas
- CHU de Quebec Universite Laval, Québec, Quebec, Canada
- Yokohama City University Medical Center, Yokohama, Japan
- Malaysia (3):
  - Hospital Wanita dan Kanak-Kanak Sabah, Kota Kinabalu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency